CLINICAL TRIAL: NCT01502527
Title: An Open Labeled Prospective Study to Investigate the Effect of Femarelle® on Vulvo-vaginal Atrophy Symptoms
Brief Title: A Twelve Week Study to Investigate the Efficacy of Femarelle®, for the Treatment of Post Menopausal Vaginal Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lila Nachtigall Rapid Medical Research, New York (Other)
Collaborators: Se-cure Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCS - 001
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Vulvo Vaginal Atrophy
Keywords: Vulvo vaginal atrophy; Femarelle
MeSH Terms: interventions — DT56a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with Femarelle (Experimental): An open labeled , twice daily treatment with Femarelle
  Interventions: Dietary Supplement: Femarelle

INTERVENTIONS:
Dietary Supplement: Femarelle — Twice daily oral treatment with Femarelle
  Other Names: DT56a

SUMMARY:
Based on previous data published on the SERM properties of Femarelle, the investigators hypothesized that Femarelle could be a potential treatment for Vulvo-vaginal atrophy(VVA) symptoms. The current study was a pilot study to examine the effect of Femarelle® on VVA symptoms in symptomatic post-menopausal women.

DETAILED DESCRIPTION:
Post-menopausal women aged 54-77, with vaginal atrophy (< 5% superficial cells on cervical cytology) with at least one moderate-to-severe VVA symptom (dryness, irritation, soreness, dysuria, dyspareunia, or bleeding with coitus), will be recruited for a 12-week open-label pilot study. The study protocol was approved by Schulman Associates IRB.Femarelle will be given twice daily and subjective symptoms as well as objective measures like inspection and vaginal pH will be measured.

ELIGIBILITY:
Inclusion Criteria:

Healthy post menopausal women between the ages of 40-85+yrs who complain of vaginal dryness with at least three urogenital symptoms from the following: vaginal dryness, vaginal irritation, vaginal soreness, dysuria, dyspareunia, bleeding with coitus & one of these symptoms must be moderate to severe as determined by patient, Moderate: discomforting and aware of it with activities. Severe: discomforting enough to interfere with activities Activities include sitting, walking, running, urinating, as well as sexual activity

* BMI 18-34 (inclusive).
* Patients having a LMP at least one year ago, either natural or surgical.
* Patients with a normal mammogram within 9 months prior to enrollment.
* Patients able to adhere to the visit schedule and protocol requirements and be available to complete the study.
* Patients who provide written informed consent to participate in the study.
* FSH > 40 mIU/m.
* Estradiol < 20 pg/ml.
* Vaginal PH > 5.
* < 5% superficial cells as assessed by vaginal cytology.
* Normal pelvic and breast exams by investigator.

Exclusion Criteria:

Patients using HRT (cannot have used for past 3 months).

* Patients consuming over the last three months high soy diet or any foods or other compounds that are sold as remedies for the post menopausal symptoms.
* Any history of significant cancer or pre-cancer, neurological, renal, cardiovascular, respiratory (e.g. asthma, COPD), hypercoagulability, hematopoietic disease, immune deficiency or any other clinically significant medical disorder, which in the investigator's judgment contraindicate administration of the study medications.
* Patients with any clinically significant abnormality upon examination at screening visit.
* Patients with a known history of drug or alcohol abuse.
* Known hypersensitivity and/or allergy to soy or flax.
* Participation in another clinical trial within the past 30 days.

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
improvement in VVA symptoms | 12 weeks
  Subjective and objective measures of VVA

CONTACTS AND LOCATIONS:
Overall Officials: Lila Nachtigall, MD, Principal Investigator — Rapid Medical Research of New York
Locations (1):
- Rapid Medical Research of New York, New York, New York, United States